CLINICAL TRIAL: NCT05834270
Title: Single Dose Versus Double Dose Tamsulosin in Management of Moderate and Severe Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: Single Dose Versus Double Dose Tamsulosin in Management of Moderate and Severe LUTS Due to BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed M. Hassan, Dr, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD vs DD Tamsulosin
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Prostatic Neoplasms; Prostate Disease; Prostate Obstruction; Prostate Hypertrophy
Keywords: Tamsulosin; Prostate
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose tamsulosin 0.4mg (Active Comparator): Single dose tamsulosin 0.4mg
  Interventions: Drug: Single dose tamsulosin 0.4mg
- Double dose tamsulosin 0.4mg (Active Comparator): Double dose tamsulosin 0.4mg
  Interventions: Drug: Double dose tamsulosin 0.4mg

INTERVENTIONS:
Drug: Single dose tamsulosin 0.4mg — Single dose tamsulosin 0.4mg
  Arms: Single dose tamsulosin 0.4mg
Drug: Double dose tamsulosin 0.4mg — Double dose tamsulosin 0.4mg
  Arms: Double dose tamsulosin 0.4mg

SUMMARY:
Single dose versus double dose tamsulosin in Management of Moderate and severe lower urinary tract symptoms due to benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* age more than 50 years
* moderate to severe lower urinary tract symptoms

Exclusion Criteria:

* prostatic cancer
* urethral stricture
* prostate surgery
* Neurogenic bladder

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the lower urinary tract symptoms | 3 months
  Assessed by the improvement in the internal prostatic symptoms score (IPSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No